CLINICAL TRIAL: NCT02469064
Title: Effects of Respiratory Muscle Training in Mechanically Ventilated Adults
Acronym: RMTMVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: Universidad del Valle, Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1755
Record Dates: First submitted 2015-06-02; First posted 2015-06-11 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Muscle Weakness
Keywords: mechanical ventilation; respiratory muscle; weaning; training; Intensive care
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Respiratory Muscle Training (Experimental): Experimental group receives as additional treatment respiratory muscle training.
  Interventions: Other: Respiratory muscle training; Other: Cardiopulmonary Physical Therapy
- Conventional physical therapy (Active Comparator): Conventional Cardiopulmonary Physical Therapy
  Interventions: Other: Cardiopulmonary Physical Therapy

INTERVENTIONS:
Other: Respiratory muscle training — Respiratory muscle training is done twice every day, with 3 series of 10 repetitions each, with a resting pause of two minutes between series (during resting time, patient is connected to mechanical ventilation again). We adjust initial load for respiratory muscle training as 50% of MIP. At the end of every training session, we assess dyspnea (perceived effort) using Modified Borg Scale (23). Four physical therapists are in charge of Respiratory muscle training, these therapists work at ICU and have experience with critically ill patients.
  Arms: Respiratory Muscle Training
Other: Cardiopulmonary Physical Therapy — Control group receives Cardiopulmonary Physical Therapy every 6 hours, physical therapy and mechanical ventilation management

SUMMARY:
Respiratory muscle training (RMT) is considered a therapeutic strategy to improve respiratory muscle strength in mechanically ventilated (MV) patients and facilitates ventilator weaning. RMT aims at improving strength and endurance of respiratory muscles . However, scarce research exists regarding evaluation of RMT in MV patients and additionally studies differ in methods, RMT protocols and subjects included. There are not reports about Colombian studies evaluating RMT effects on MV patients. The aim of this study is to evaluate the effectiveness of respiratory muscle training in increasing respiratory muscle strength and improving weaning outcomes in MV patients who required ventilatory support for more than 48 hours at an Intensive Care Unit of an IV level Hospital in Cali during the period 2014-2015

DETAILED DESCRIPTION:
Patients who have been under mechanical ventilation for 48 hours are invited for participation in this study. Once participants are identified and his/her legal representative has decided to participate through an informed consent, subjects are randomly assigned to the experimental or conventional group.

Data collection begins with registering individual information into a data collection form that has been designed for the study; muscle strength is measured as Maximum Inspiratory Pressure (MIP). Then, patients are assigned either to experimental or group control using opaque sealed envelopes. Stratified randomization is performed, using SEPSIS status as strata, and within each category randomization block size is 4 and 6 respectively. Once sepsis status has been established, green envelopes are opened for patients with sepsis, and blue envelopes are opened for patients without sepsis. Finally intervention is performed according to group assignment.

Interventions

Conventional Therapy Group Control group receives conventional intervention of Cardiopulmonary Physical Therapy which has been established by institutional protocols, and consists of Cardiopulmonary Physical Therapy every 6 hours, physical therapy and mechanical ventilation management

Measuring Respiratory Muscle Strength

Respiratory muscle strength is measured by Maximum inspiratory pressure (MIP) following American Thoracic Society (ATS) and European Respiratory Society (ERS). protocols. MIP measures are performed in both groups, experimental and control. To measure MIP, we ask the patient to do a maximum inspiration and then hold it for 5 seconds; this inspiration begins from functional residual capacity (FRC). We will perform 3 measures with each patient and register the highest value obtained, using a Manuvacuometer for this measure.

Experimental Group

The experimental group will receive conventional treatment plus a respiratory muscle training protocol. Respiratory muscle training utilizes a Threshold device (IMT from Respironics Inc;Murrysville, USA), this device has been validated both in healthy subjects and in chronic obstructive pulmonary disease (COPD) patients

Study Setting

This study is being conducted at the Adult Intensive Care Unit in Valle del Lili Foundation, a private health institution level IV, located in the south of Cali, this is a referral centre for the southwest of Colombia.

Data Collection

Instrument design and pilot study

The researchers designed data collection tool to register data from clinical records and intervention, this tool is being used for both groups. The data collection tool includes demographic, clinical and intervention variables.

A pilot trial in a group of patients with similar characteristics to the study sample was conducted and then some aspects of the data collection tool and measuring protocols were adjusted

Research team and field personnel training

Four physical therapy specialists who had more than 4 years of experience in intensive care were recruited as monitors and data collectors.

In order to standardise and to determine validity of MIP measuring protocol, principal researcher conducted a training session with the physical therapists and then intra and inter-rater validity in 30 healthy subjects was established.

The primary source of information was the data collection tool, which was filed during intervention with each subject. The secondary source of information is the electronic medical record, recorded data are reliable because they are a basis for decision making in critically ill patients.

Patient recruiting and monitoring is performed by four physical therapists mentioned before. Data collection occurs from Monday to Sunday between 8:00 a.m. to 6:00 pm. Main researcher is not involved in data collection or intervention.

The variables obtained on patient admission to the study are: type of intervention, age, gender, medical history, diagnosis at admission, Severity Index (Apache II), hours of mechanical ventilation, weaning hours, cumulative dose of sedative received, cumulative dose of analgesics received, cumulative dose of relaxant received, cumulative dose of steroids, socioeconomic status and educational level.

The variable obtained during follow-up is: respiratory muscle strength.

The variables obtained at the end of follow-up are: Number of sessions of respiratory muscle training received, mechanical ventilation time (in hours), total hours of weaning, cumulative dose of sedatives, cumulative dose of pain medication received, cumulative dose of steroids, received physical therapy, number of physical therapy sessions, pulmonary rehabilitation received, number of pulmonary rehabilitation sessions, Non Invasive Ventilation requirement, pulmonary rehabilitation number of sessions, death, reintubation requirement, reintubation date, number of extubated hours because of reintubation, tracheotomy, tracheotomy date, septic shock, date of septic shock, death, date of death, decision not to continue in the study (date).

Data Quality

A monthly checking of data collection tools is performed by the principal investigator, using a checklist and comparing data recorded in the tool with medical records of subjects, this procedure is done before transcribing information on to the study database. Additionally, every data collection tool is reviewed using a checklist that includes three quality indicators: days between follow-up completion and closing of tool, number of empty boxes, number of diagnoses that are inconsistent; this procedure is also a responsibility for the principal investigator. Monthly meetings with the study team are held to talk about recording faults and how to improve quality of data collection and registration.

Database design and management

Once the data in the data collection tools have been checked, information is registered in an Epi Info database and then this will be exported to STATA 12 for analysis. Data registering in the Epi Info database will be done after every data collection tool has been closed and checked by the main researcher. Data registering will be performed by a person hired and trained for these procedures. Database management and analysis is performed by the principal researcher.

Data Analysis Plan

Patient recruitment and following-up are described using a flowchart designed according to CONSORT statement 2010. A preliminary exploratory data analysis will be conducted to evaluate data performance and basic assumptions required to implement statistical tests (normality, linearity and homoscedasticity). This analysis will also allow us to identify errors and biases in data collected, as well as outliers and missing data.

Sociodemographic and clinical characteristics of patients at study entry will be analysed descriptively according to measurement level of every variable using central tendency, dispersion measures, frequency tables and 95% confidence intervals. An analysis of clinical and sociodemographic characteristics of eligible patients who met inclusion criteria but were not included in the study will also be performed, as well as the reasons for not being included; this analysis will allow us to identify selection bias.

Finally univariate and multivariate analysis will be performed according to study objectives. Analysis will be performed on an intention to treat basis for all patients.

Respiratory Muscle Strength (MIP): Presuming that there is data normality, at univariate analysis, a difference between final MIP means of experimental group and control group will be analysed using a t-student. Differences in MIP means within every group will be analysed using linear regression. If normality, error independency and homoscedasticity are not met, we will consider data transformation for MIP variables. Once linear regression is performed a diagnostic test will be done to evaluate if the model represents or mimic observed data. In order to control for potential confusing factor an adjustment of variables will be done, we are considering as confusing factors: i)Cumulative medicament doses received before intervention, ii)Cumulative medicament doses received, iii) Time in ventilation mode before intervention, iv)Time in every ventilatory mode during intervention, v) Admission diagnoses. Additionally we will evaluate effect modification between variables mentioned before.

Ventilation time and weaning time: we will perform univariate analysis of total weaning time and total ventilation time between experimental and control group using a survival analysis (Kaplan-Meyer). We also intend to do multivariate analysis of total weaning time and total ventilation time using Cox regression adjusting potential confusing factors that we considered with other variables. We will verify Cox model assumptions about hazard proportionality during following-up. Need for reintubation: We are doing univariate analysis of need for reintubation using a comparison of proportions with Chi-square or Fischer exact test. Need for reintubation Relative Risk (RR) will also be determined for patients in both groups (Control and Experimental). We are doing multivariate analysis for the need for reintubation with logistic regression adjusting for potential confusing factors mentioned before.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years at least
* Informed consent to participate in study by legal representative or family member
* First event requiring mechanical ventilation
* Being intubated at the study setting ( Valle del Lili Foundation) or at peripheral services and referred 12 hours or less after intubation
* Adequate gas interchange: Blood pressure of oxygen > 60 mmHg with Inspired fraction of oxygen ≤ 0. 5 and positive pressure at end of expiration (PEEP) < 8 cmh20
* Sedation level between -1 and 0 (24, 25)
* Hemodynamic stability: Medium arterial blood pressure > 60 mmHg without vasopressors or requiring a minimum of vasopressor support (epinephrine < 0,4 mcg/Kg/ min)

Exclusion Criteria:

* Progressive neuromuscular disease such as Amyotrophic Lateral Sclerosis , Muscular Dystrophy, Multiple Sclerosis, Myasthenia Gravis, or other neuromuscular disorder that could interfere with response to inspiratory muscle training .
* Central nervous system disorders: severe traumatic brain injury
* Spinal cord injury at a level higher than T8
* Chest or spine skeletal disorders (scoliosis, flail chest, spine surgery) that limit movement of ribs and rib cage.
* Requirement of ventilatory support at home prior to hospitalization
* Presence of excessive secretions (requiring more than one suctioning procedure every hour).
* Tracheostomy
* Previous requirement of mechanical ventilation during this period of hospitalization
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lina M Sandoval, PT, Principal Investigator — Fundacion Valle del Lili- Universidad del Valle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346
- [Background] Sprague SS, Hopkins PD. Use of inspiratory strength training to wean six patients who were ventilator-dependent. Phys Ther. 2003 Feb;83(2):171-81. PMID 12564952
- [Background] Martin AD, Davenport PD, Franceschi AC, Harman E. Use of inspiratory muscle strength training to facilitate ventilator weaning: a series of 10 consecutive patients. Chest. 2002 Jul;122(1):192-6. doi: 10.1378/chest.122.1.192. PMID 12114357
- [Background] Caruso P, Denari SD, Ruiz SA, Bernal KG, Manfrin GM, Friedrich C, Deheinzelin D. Inspiratory muscle training is ineffective in mechanically ventilated critically ill patients. Clinics (Sao Paulo). 2005 Dec;60(6):479-84. doi: 10.1590/s1807-59322005000600009. Epub 2005 Dec 12. PMID 16358138
- [Background] Bissett B, Leditschke IA, Green M. Specific inspiratory muscle training is safe in selected patients who are ventilator-dependent: a case series. Intensive Crit Care Nurs. 2012 Apr;28(2):98-104. doi: 10.1016/j.iccn.2012.01.003. Epub 2012 Feb 15. PMID 22340987
- [Background] Bissett B, Leditschke IA. Inspiratory muscle training to enhance weaning from mechanical ventilation. Anaesth Intensive Care. 2007 Oct;35(5):776-9. doi: 10.1177/0310057X0703500520. PMID 17933168
- [Background] Chang AT, Boots RJ, Henderson R, Paratz JD, Hodges PW. Case report: inspiratory muscle training in chronic critically ill patients--a report of two cases. Physiother Res Int. 2005;10(4):222-6. doi: 10.1002/pri.14. PMID 16411617
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Cader SA, Vale RG, Castro JC, Bacelar SC, Biehl C, Gomes MC, Cabrer WE, Dantas EH. Inspiratory muscle training improves maximal inspiratory pressure and may assist weaning in older intubated patients: a randomised trial. J Physiother. 2010;56(3):171-7. doi: 10.1016/s1836-9553(10)70022-9. PMID 20795923
- [Background] Chang AT, Boots RJ, Brown MG, Paratz J, Hodges PW. Reduced inspiratory muscle endurance following successful weaning from prolonged mechanical ventilation. Chest. 2005 Aug;128(2):553-9. doi: 10.1378/chest.128.2.553. PMID 16100137
- [Background] Condessa RL, Brauner JS, Saul AL, Baptista M, Silva AC, Vieira SR. Inspiratory muscle training did not accelerate weaning from mechanical ventilation but did improve tidal volume and maximal respiratory pressures: a randomised trial. J Physiother. 2013 Jun;59(2):101-7. doi: 10.1016/S1836-9553(13)70162-0. PMID 23663795
- [Derived] Sandoval Moreno LM, Casas Quiroga IC, Wilches Luna EC, Garcia AF. Efficacy of respiratory muscle training in weaning of mechanical ventilation in patients with mechanical ventilation for 48hours or more: A Randomized Controlled Clinical Trial. Med Intensiva (Engl Ed). 2019 Mar;43(2):79-89. doi: 10.1016/j.medin.2017.11.010. Epub 2018 Feb 3. English, Spanish. PMID 29398169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted seven months. The collection was performed in an Intensive Care Unit of a IV level clinic in the city of Cali
Pre-assignment Details: 126 patients were randomized, 3 of them did not comply with the protocol, being assigned to the experimental treatment and receiving conventional treatment.
  No patient requested to be withdrawn from the study, and no patient had any adverse effects
Groups:
- Respiratory Muscle Training: Experimental group receives as additional treatment respiratory muscle training.
  Respiratory muscle training: Respiratory muscle training is done twice every day, with 3 series of 10 repetitions each, with a resting pause of two minutes between series (during resting time, patient is connected to mechanical ventilation again). We adjust initial load for respiratory muscle training as 50% of maximum inspiratory pressure (MIP). At the end of every training session, we assess dyspnea (perceived effort) using Modified Borg Scale (23). Four physical therapists are in charge of Respiratory muscle training, these therapists work at intensive care unit (ICU) and have experience with critically ill patients.
  Cardiopulmonary Physical Therapy: Control group receives Cardiopulmonary Physical Therapy every 6 hours, physical therapy and mechanical ventilation management
Period: Overall Study
Arm/Group | Conventional Physical Therapy | Respiratory Muscle Training
Started | 64 | 62
Completed | 63 | 59
Not Completed | 1 | 3
Not completed — Request not to receive intervention. | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Respiratory Muscle Training | Conventional Physical Therapy | Total
Number analyzed (Participants) | 62 | 64 | 126
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [40 to 70] | 64 [47 to 72] | 62 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 33 | 38 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 62 | 64 | 126

OUTCOME MEASURES:

1. Primary Outcome: Weaning Time From Mechanical Ventilation
Description: Weaning time was considered as time elapsed from beginning of pressure support mode in mechanical ventilation (Pressure support at 10 centimeters of water (cmsH2O) or less) or continuous positive pressure in the airway mode (CPAP) until patient extubation
Time Frame: Measured by the end of the period of mechanical ventilation, an average expected time of 4 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Respiratory Muscle Training | Conventional Physical Therapy
Number analyzed (Participants) | 62 | 64
hours | 5 [0 to 72] | 5 [0 to 59]
Statistical Analysis 1: Comparison: Respiratory Muscle Training vs Conventional Physical Therapy; Test type: Other; p = 0.84, Mann Whitneey; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.55 to 1.20] — Univariate analysis of the probability of extubation was performed using Kaplan-Meir survival analysis and the logrank test.The multivariate analysis was performed by cox regression, a simple model was performed and a final model

2. Secondary Outcome: Changes in Maximum Inspiratory Pressure (MIP)
Description: Changes in Maximum Inspiratory Pressure (MIP) was considered as Final MIP minus baseline MIP
Time Frame: Measured at baseline (baseline MIP) and right before patient extubation (finalMIP, an average of 2 hours)
Population: 24 patients did not reach a measurement of the Final MIP, of them, 14 belonged to the experimental treatment group and 10 to the conventional treatment group; therefore this result was analyzed in 102 patients.
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Respiratory Muscle Training | Conventional Physical Therapy
Number analyzed (Participants) | 48 | 54
cmH20 | 9.43 (17.48) | 5.92 (3.51)
Statistical Analysis 1: Comparison: Respiratory Muscle Training vs Conventional Physical Therapy; Test type: Other; p = 0.48, t-test, 2 sided; Slope = 0.46, 95% CI 2-sided [-3.75 to 4.78] — The slope shows the difference between the means of the change in the MIP of the group that received the experimental treatment and the group that received the conventional treatment

ADVERSE EVENTS:
Time Frame: The search for adverse events was performed up to 48 hours after the patients reached the end point of follow-up.
Description: The search for adverse events was performed daily by two physiotherapists who were part of the field work, by an institutional doctor who is part of the ICU team external to the work and by the coordinator of the respiratory therapy group. In order to search for adverse events, the Standardized Operational Manual Adverse Event Reporting was designed and the adverse events that are most likely to occur in this population extracted from the Common Terminology for Adverse Events
Arm/Group | Respiratory Muscle Training | Conventional Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 0/62 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No